CLINICAL TRIAL: NCT06494202
Title: Stroke Rehabilitation: A Systemized and Hierarchized Rehabilitation Program for the Brazilian Unified Health System
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Collaborators: Ministry of Health, Brazil (Other Government)
Responsible Party: Principal Investigator, Marta Imamura, MD, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 78062224.5.0000.0068
Record Dates: First submitted 2024-07-02; First posted 2024-07-10 (Actual); Last update posted 2024-07-31 (Actual); Status verified 2024-07

CONDITIONS: Stroke, Ischemic
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Masking Description: Different collaborators will be care providers and outcomes assessors.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional rehabilitation program (Active Comparator): Conventional rehabilitation intervention with multidisciplinary team (medical services, physiotherapy, occupational therapy, physical education, psychology, nutrition, social service, speech therapy, and nurse) delivered during four to six weeks of intensive in-patient program
  Interventions: Other: Conventional rehabilitation program.
- Innovative rehabilitation program (Experimental): Conventional rehabilitation intervention with multidisciplinary team (medical services, physiotherapy, occupational therapy, physical education, psychology, nutrition, social service, speech therapy, and nurse) delivered during four to six weeks of intensive in-patient program combined with innovative medical therapies (laser therapy, radial extracorporeal shockwaves therapy, focused extracorporeal shockwaves therapy, segmentary desensibilization with lidocaine, functional electrical stimulation - FES).
  Interventions: Other: Innovative rehabilitation; Other: Conventional rehabilitation program.

INTERVENTIONS:
Other: Innovative rehabilitation — Conventional rehabilitation program associated with innovative therapies.
  Arms: Innovative rehabilitation program
Other: Conventional rehabilitation program. — Conventional rehabilitation program

SUMMARY:
The goal of this clinical trial is to systemize and hierarchize a rehabilitation program for the Brazilian Unified Health System in patients with stroke above 18 years of age and of both sexes. The main question it aims to answer is:

* Do patients with ischemic first episode of stroke have central nervous systems consequences due to peripheral and central nervous system sensibilization?
* Can stroke patients benefit from a systemized and hierarchized rehabilitation program with desensibilization interventions combined with multidisciplinary and educational programs?

We will randomize 60 patients, 30 in each study arm.

Researchers will compare the intervention group with an active control whose treatment is the institutional conventional program to see if innovative desensibilization strategies yield superior results. Authors will also investigate the role of genetic polymorphism and ancestrality in the outcome measures.

Participants will undertake an innovative or conventional rehabilitation program, according to the randomization.

ELIGIBILITY:
Inclusion Criteria:

* Clinical and radiological (magnetic resonance or tomography) diagnosis of ischemic stroke;
* Single episode of stroke;
* Clinical stability according to medical assessment;
* Time since stroke onset no longer than 24 months;
* Capacity to understand the study procedures;
* Eligible to be admitted to hospitalization at the institute where the study will be conducted
* Agree to sign the Informed Consent Form (ICF).

Exclusion Criteria:

* Presence of psychiatric disorders;
* Presence of subarachnoid hemorrhage;
* Presence of intracerebral hemorrhage;
* Presence of neuromuscular disorders;
* Presence of other neurological diseases or brain neoplasm;
* Presence of cognitive disorders measured with Montreal Cognitive Assessment (MoCA), scores below 20 points;
* Presence of systemic arterial hypertension (systolic blood pressure ≥ 185mmHg or diastolic blood pressure ≥ 110 mmHg).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-10-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Motor recovery | Change from baseline to six weeks of intervention.
  Motor recovery measured with Fugl-Meyer Assessment (FMA), ranging from 0 to 100 for upper and lower extremities combined. Higher scores mean better outcome.

SECONDARY OUTCOMES:
Functional independence | Change from baseline to six weeks of intervention.
  Functional independence measured with Functional Independence Measure (FIM). This scale ranges from 18 to 126, and higher scores mean better outcomes.
Muscle strength | Change from baseline to six weeks of intervention.
  Muscle strength measured Medical Research Council scale (MRC). The MRC is a scale that ranges from 0 to 5 and higher scores mean better outcomes.
Upper extremity recovery | Change from baseline to six weeks of intervention.
  Finger movement measured with Finger Tapping assessement. The finger tapping assessment measures the number index finger movements (up and down) performed for one minute.
Spasticity reduction | Change from baseline to six weeks of intervention.
  Upper limbs spasticity measured with Modified Ashworth Scale (MAS). The MAS ranges from 0 to 4, and higher scores mean worse outcomes.
Gait recovery | Change from baseline to six weeks of intervention.
  Gait recovery measured with 10-meter walk test (10mwt).
Gait and balance recovery | Change from baseline to six weeks of intervention.
  Gait and balance recovery measured with Timed Up and Go (TUG).
Pain assessment | Change from baseline to six weeks of intervention.
  Pain intensity measured with Visual Analogue Scale (VAS). The VAS is a linear approximation of pain intensity ranging from 0 to 10 and higher scores mean worse outcomes.
Quality of life after stroke | Change from baseline to six weeks of intervention.
  Quality of Life after stroke measured with Stroke Impact Scale (SIS). The SIS ranges from 0 to 100 and higher scores mean better outcomes.
Sensibilization assessment | Change from baseline to six weeks of intervention.
  Sensibilization assessment conducted with Pain Pressure Threshold (PPT).

OTHER OUTCOMES:
Physical Activity | Baseline.
  Level of physical activity measured with 3-D accelerometer (ActigraphwGT3x-BT ).
Postural control | Change from baseline to six weeks of intervention.
  Postural control measured with pressure platforms combined with static activities and cognitive activities.
Nutritional status | Baseline.
  Nutritional status described with nutrition questionnaire. The questionnaire ranges from 0 to 100 and higher scores mean better outcomes.
Body Mass Index (BMI) | Baseline
  BMI measured with weight and height and the widely known formula.
Stool assessment | Baseline
  Stool classification based on Bristol Stool Scale. This scale classifies the feces into seven Types. Types 3 and 4 indicate good better outcomes and the extremities of this classification indicate worse outcomes.
Excessive daytime sleepiness | Change from baseline to six weeks of intervention.
  Excessive daytime sleepiness measured with Epworth Sleepiness Scale. This scale ranges from 0 to 24 and higher scores mean worse outcome.
Sleep quality assessment - Questionnaire | Change from baseline to six weeks of intervention.
  Sleep quality measured with Pittsburgh Sleep Quality Index. This is a scale that ranges from 0 to 21 and higher scores indicate worse outcome.
Sleep quality assessment - digital assessment | Change from baseline to six weeks of intervention.
  Sleep quality measured with digital actigraphy.
Physical activity | Change from baseline to six weeks of intervention.
  Physical activity fitness tested with exercise bike.
Handgrip strength | Change from baseline to six weeks of intervention.
  Handgrip strength measured with dynamometer.
Sarcopenia | Baseline
  Sarcopenia determined with a combination of handgrip strength, sit-to-stand, and ultrasonography.
Lower limb muscle strength | Baseline
  Lower limb muscle strength measured with Sit-to-stand test.
Muscle thickness | Baseline
  Lower limb muscle thickness assessed with ultrasound of the vastus intermedius muscle.
Ancestrality | Baseline.
  Role of ancestrality in the outcome measures. A blood sample will be used for this outcome.
Genetic polymorphisms | Baseline.
  Role of genetic polymorphism the outcome measures. A blood sample will be used for this outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Marta Imamura, Professor, Principal Investigator — Instituto de Medicina Física e Reabilitação - FMUSP
Locations (1):
- Instituto de Medicina Física e Reabilitação (IMREA-FMUSP), São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Yes
Study data will be made available under reasonable request after publication. Data will include de-identified participant data and the data dictionary. Requests can be submitted to the corresponding author. Request will be analyzed and ethical and legal implications of data sharing will be considered. Data will be shared after consent of study participants
  Brazil is under Brazilian General Data Protection Law (LGPD, English translation) and all shared data will require participants prior consent.
Time Frame: After publication under reasonable request.
Access Criteria: Reasonable request and participants prior consent.